CLINICAL TRIAL: NCT00106080
Title: Improving the Quality of End-of-Life Communication for Patients With COPD
Brief Title: Improving the Quality of End-of-Life Communication for Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IIR 02-292
Record Dates: First submitted 2005-03-18; First posted 2005-03-21 (Estimated); Results first posted 2014-11-11 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Pulmonary Disease; COPD; Chronic Bronchitis; Emphysema
Keywords: Communication; Palliative Care
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema; Communication

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Audit and Feedback
  Interventions: Behavioral: Audit and Feedback
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Audit and Feedback — Intervention patients and clinicians received a one-page patient-specific individualized summary, based on questionnaire responses, to stimulate conversations.
  Arms: Intervention

SUMMARY:
The purpose of this study is to evaluate a multifaceted intervention to improve the quality of end-of-life communication between patients with COPD and their primary care providers using information about patients preferences for end of life care and how to communicate and use this information to activate patients, family members, and healthcare providers.

DETAILED DESCRIPTION:
This project builds on previous work that described preferences important to patients at end-of-life and desire for life-sustaining therapy by incorporating these attributes into a multifaceted intervention designed to improve the quality of end-of-life communication.

Our specific aim was to evaluate a multifaceted intervention to improve the quality of end-of-life communication between patients with moderate or severe COPD and their primary care providers. The intervention is based on self-efficacy theory and includes provider education, local champions and role models, determination of patients individual barriers and facilitators regarding communication about end-of-life care, preferences for communication about end-of-life care and preferences for end-of-life care and using this information to activate patients, family members, and healthcare providers.

For both control and intervention patients we collected the following information which was incorporated into a one-page summary report:

1. Preferences about cardiopulmonary resuscitation (CPR) and mechanical ventilation
2. Preferences for communication with provider
3. Measure of severity of airflow obstruction
4. Barriers and facilitators to communication
5. Preferences for end-of-life care

The intervention was incorporated into a usual clinic visit. For the upcoming clinic visit, we generated an individualized one-page patient specific feedback form for intervention group patients and providers. Patients and providers in the control group did not receive the form.

The generated one-page feedback form was:

1. Mailed to the patient to share with their surrogate
2. Sent to their provider prior to the clinic visit
3. Provided to the patient prior to their clinic visit

The methods used for this study could be translated into clinic practice and possibly generalized to other chronic life-threatening conditions.

ELIGIBILITY:
Inclusion Criteria:

One or more of the following:

1 Have 3 or more outpatient clinics visits for COPD (ICD-9) in the two years prior to enrollment.

2. Have been hospitalized with a primary discharge diagnosis (ICD-9) for COPD in the two years prior to enrollment.

3. Active use of inhaled beta-agonist and ipratropium bromide (or equivalent in combination inhalers like Combivent) in the 12 months prior to enrollment.

Plus

1. Have a future visit scheduled in one of the eligible primary care or chest clinics; and
2. Have airflow limitation

Exclusion Criteria:

1. If they have cognitive dysfunction, language barriers or severe psychiatric disorder that would preclude them from completing the questionnaires. This was assessed initially by the patients provider and by the research assistant during in-person interviews.
2. The provider taking care of their COPD does not participate.
3. Have a new diagnosis of COPD within the last month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2004-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Au, MD MS, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

REFERENCES:
- [Result] Curtis JR, Engelberg RA, Wenrich MD, Au DH. Communication about palliative care for patients with chronic obstructive pulmonary disease. J Palliat Care. 2005 Autumn;21(3):157-64. PMID 16334970
- [Result] Reinke LF, Slatore CG, Udris EM, Moss BR, Johnson EA, Au DH. The association of depression and preferences for life-sustaining treatments in veterans with chronic obstructive pulmonary disease. J Pain Symptom Manage. 2011 Feb;41(2):402-11. doi: 10.1016/j.jpainsymman.2010.05.012. Epub 2010 Dec 8. PMID 21145201
- [Result] Janssen DJ, Curtis JR, Au DH, Spruit MA, Downey L, Schols JM, Wouters EF, Engelberg RA. Patient-clinician communication about end-of-life care for Dutch and US patients with COPD. Eur Respir J. 2011 Aug;38(2):268-76. doi: 10.1183/09031936.00157710. Epub 2011 Jan 13. PMID 21233263
- [Result] Cecere LM, Slatore CG, Uman JE, Evans LE, Udris EM, Bryson CL, Au DH. Adherence to long-acting inhaled therapies among patients with chronic obstructive pulmonary disease (COPD). COPD. 2012 Jun;9(3):251-8. doi: 10.3109/15412555.2011.650241. Epub 2012 Apr 12. PMID 22497533
- [Result] Cecere LM, Littman AJ, Slatore CG, Udris EM, Bryson CL, Boyko EJ, Pierson DJ, Au DH. Obesity and COPD: associated symptoms, health-related quality of life, and medication use. COPD. 2011 Aug;8(4):275-84. doi: 10.3109/15412555.2011.586660. Epub 2011 Aug 2. PMID 21809909
- [Result] Au DH, Udris EM, Engelberg RA, Diehr PH, Bryson CL, Reinke LF, Curtis JR. A randomized trial to improve communication about end-of-life care among patients with COPD. Chest. 2012 Mar;141(3):726-735. doi: 10.1378/chest.11-0362. Epub 2011 Sep 22. PMID 21940765
- [Result] Reinke LF, Slatore CG, Uman J, Udris EM, Moss BR, Engelberg RA, Au DH. Patient-clinician communication about end-of-life care topics: is anyone talking to patients with chronic obstructive pulmonary disease? J Palliat Med. 2011 Aug;14(8):923-8. doi: 10.1089/jpm.2010.0509. Epub 2011 Jun 1. PMID 21631367
- [Result] Reinke LF, Uman J, Udris EM, Moss BR, Au DH. Preferences for death and dying among veterans with chronic obstructive pulmonary disease. Am J Hosp Palliat Care. 2013 Dec;30(8):768-72. doi: 10.1177/1049909112471579. Epub 2013 Jan 8. PMID 23298873

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients gave written informed consent before enrollment.
Groups:
- Intervention (Audit and Feedback): We solicited patients' preferences for health care communication and treatment in order to generate individualized summary reports of patient's preferences. These individualized summaries of patient's preferences regarding communication about end-of-life care and preferences for end-of-life care were used to activate patients, family members, and healthcare providers.
- Control (Usual Care): We solicited control patients' preferences but did not deliver study generated summary reports to patients, surrogates or providers.
Period: Overall Study
Arm/Group | Intervention (Audit and Feedback) | Control (Usual Care)
Started | 194 | 182
Completed | 151 | 155
Not Completed | 43 | 27
Not completed — Withdrew/Loss to follow-up | 43 | 27

BASELINE CHARACTERISTICS:
Population: 42 clinicians were randomized to the intervention group. 50 clinicians were randomized to the control group. 376 patients were enrolled and assigned to their clinician's treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 194 | 182 | 376
Age, Continuous [Mean (Standard Deviation); unit: years] — Patient age in years
  years | 69.4 (10.0) | 69.4 (10.0) | 69.4 (10.0)
Sex/Gender, Customized [Number; unit: percent] — Patient gender reported as percent.
  percent
    Male | 97.9 | 96.2 | 97.1
Race/Ethnicity, Customized [Number; unit: percent] — Patient race reported as percent.
  percent
    White | 85.3 | 87.0 | 86.1
Smoking Status [Number; unit: percent] — Patient smoking status reported as percent.
  percent
    Never smoked | 3.9 | 3.1 | 3.5
    Past smoker | 73.2 | 65.0 | 69.2
    Current smoker | 22.9 | 31.9 | 27.3
Male Clinicians [Number; unit: percent] — Clinician gender reported as percent.
  percent | 50.0 | 44.0 | 47.1
Clinician clinic [Number; unit: percent] — Clinician clinic reported as percent.
  percent
    Geriatric | 7.1 | 8.0 | 7.6
    Primary care/internal medicine | 64.3 | 68.0 | 66.1
    Pulmonary | 28.6 | 24.0 | 26.4

OUTCOME MEASURES:

1. Primary Outcome: Effect of Intervention on Quality of Patient Clinician Communication About End-of-Life Care(QOC) Scale
Description: The quality of end-of-life communication (QOC) score ranges between 0 and 100, with higher scores indicating better communication between patients and providers.
Time Frame: Measured at enrollment and 2 weeks after targeted clinic visit
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 194 | 182
units on a scale
  Pre-visit | 23.3 [19.9 to 26.8] | 19.2 [15.9 to 22.4]
  Post-visit | 34.0 [28.5 to 39.4] | 25.5 [20.4 to 30.5]
Statistical Analysis 1: Comparison: Intervention vs Control; Power calculation: With 60 providers in each group, maintaining the probability of a type I error of 0.05, power of 0.90, provider level mean QOC score of 54.5 and provider level standard deviation in QOC score of 12.0, the minimal detectable difference in QOC score would be 7.5; Test type: Superiority or Other; p = 0.03, GEE regression — No multiple comparisons, a priori threshold < 0.05; Generalized estimating equations (GEE) regression, clustering for provider; Difference between groups after adjust = 5.7

2. Secondary Outcome: Effect of Intervention on Patient Reported Discussions About Treatment Preferences at Their Last Clinic Visit.
Description: We measured the difference between intervention and control group patients reporting having had a discussion with their clinician about treatment preferences at their last clinic visit.
Time Frame: Assessed 2 weeks after targeted clinic visit
Measure: Number (95% Confidence Interval); unit: Proportion of participants reporting
Arm/Group | Intervention | Control
Number analyzed (Participants) | 194 | 182
Proportion of participants reporting | 0.30 [0.19 to 0.41] | 0.11 [0.06 to 0.16]

ADVERSE EVENTS:
Arm/Group | Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/194 | 0/182
Other Adverse Events (participants affected / at risk) | 0/194 | 0/182

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Informed Consent Form (2007-07-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT00106080/ICF_000.pdf